CLINICAL TRIAL: NCT03601871
Title: The Efficacy and Safety of Thalidomide in Preventing Multi-cycle, Cisplatin-containing CINV: a Pragmatic Randomized Open-label Clinical Trial
Brief Title: The Efficacy and Safety of Thalidomide in Preventing CINV Induced by Cisplatin-containing Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yunpeng Liu (Other)
Responsible Party: Sponsor-Investigator, Yunpeng Liu, Director of Department of Medical Oncology，The First Hospital of China Medical University, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CLOG1801
Record Dates: First submitted 2018-05-30; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Thalidomide; Chemotherapy-induced Nausea and Vomiting; cisplatin
MeSH Terms: conditions — Vomiting | interventions — Thalidomide; Dexamethasone; Serotonin 5-HT3 Receptor Antagonists; Palonosetron

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Palonosetron 0.25 mg intravenously on day 1; or 1st-generation 5-HT3 antagonists (used as clinal routine) on day 1-3; Dexamethasone 12 mg by mouth or intravenously before chemotherapy on day 1 and 8 mg on days 2-4.
  Interventions: Drug: Dexamethasone; Drug: 5-HT3 antagonists
- Thalidomide group (Experimental): Thalidomide 100 mg by mouth twice a day on days 1-5; Palonosetron 0.25 mg intravenously on day 1; or 1st-generation 5-HT3 antagonists (used as clinal routine) on day 1-3; Dexamethasone 12 mg by mouth or intravenously before chemotherapy on day 1 and 8 mg on days 2-4.
  Interventions: Drug: Thalidomide; Drug: Dexamethasone; Drug: 5-HT3 antagonists

INTERVENTIONS:
Drug: Thalidomide — Thalidomide (Thalidomide Oral Product)100 mg by mouth twice a day on days 1-5 after chemotherapy .
  Arms: Thalidomide group
Drug: Dexamethasone — Dexamethasone 12 mg by mouth or intravenously before chemotherapy on day 1 and 8 mg on days 2-4
Drug: 5-HT3 antagonists — Palonosetron 0.25 mg intravenously on day 1; or 1st-generation 5-HT3 antagonists (used as clinal routine) on day 1-3
  Other Names: Palonosetron, or 1st-generation 5-HT3 antagonists

SUMMARY:
This is a pragmatic randomized, multi-center, open-label randomized clinical trial, aimed to evaluate efficacy and safety of thalidomide in improving prevention of chemotherapy-induced delayed nausea and vomiting (CINV) in chemotherapy-naive patients after multi-cycle cisplatin-containing highly emetogenic chemotherapy (HEC) .

DETAILED DESCRIPTION:
This is a pragmatic randomized, multi-center, open-label randomized clinical trial, aimed to evaluate efficacy and safety of thalidomide in improving prevention of chemotherapy-induced delayed nausea and vomiting (CINV) in chemotherapy-naive patients after multi-cycle cisplatin-containing highly emetogenic chemotherapy (HEC) . A total of 880 patients are planned to be enrolled into the study. Chemotherapy-naïve patients treated with multi-cycle cisplatin-containing chemotherapy will be randomized into two groups(thalidomide group and control group), and be treated with Thalidomide+5-hydroxytryptamine receptor(5-HT3) antagonist +Dexamethasone (Thalidomide group) or 5-HT3 antagonist + Dexamethasone(control group), respectively. The primary end point is no nausea rate in delayed phase of the first cycle chemotherapy, and the secondary end points include the complete response rate of vomiting in acute,delayed and overall period; no nausea rate in acute and overall phase; anorexia score, fatigue score and sedation score assessed by VAS ; safety and quality of life (QOL) during multi-cycle chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18y ≤Age≤70y
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Histologically confirmed solid neoplasm
* No prior chemotherapy
* Laboratory test must meet the following criteria: hemoglobin (HGB) ≥90g/ L, neutrophil count ≥1.5×109/L, platelet count ≥85×109/L, creatinine clearance rate (CCr) ≥60ml/min, total bilirubin (TBil) ≤1.5 upper normal limitation (UNL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 UNL (For patients with liver metastasis, the AST/ALT must be ≤5.0 UNL), blood glucose ≤11.1 mmol/L
* Life expectancy of at least 12 weeks
* Signed informed consent
* For women with child bearing potential, a negative serum or urine pregnancy test result should be obtained before enrollment;the patients and their couples should receive contraception for at least 3 years after their last dosage of thalidomide.
* Cancer patients scheduled to receive chemotherapy containing a 50 mg/m2 or higher dose of cisplatin for 4-6 cycles

Exclusion Criteria:

* Diabetic patients
* Pregnant or lactated women
* Patient with history of severe thrombosis
* Concomitant radiotherapy
* Known hypersensitivity yo thalidomide, palonosetron, or dexamethasone.
* Concurrent administration of any other drug which affect antiemetic effect evaluation such as proton pump inhibitor, H2 blocker, amifostine, sedative drugs
* Cyclophosphamide, hydroxydaunomycin, Oncovin, and prednisone (CHOP )regiment or taxanes-based regiment
* Existing emesis within 24 hours before chemotherapy administration
* Symptomatic brain metastasis or suspected clinical brain metastasis
* Serious uncontrolled systemic illness or medical condition: congestive heart failure, unstable angina, history of documented myocardial infarction within 6 months, uncontrolled hypertension and high risk uncontrollable arrhythmias; Obvious neurological or mental abnormalities including mental disorder, epileptic dementia, which affect compliance; Uncontrolled acute infections; Uncontrolled peptic ulcer or other contraindication for corticosteroid therapy.
* Inability to take or absorb oral medicine
* Concurrent administration of any other investigational drug, or have been enrolled in other clinical trial with investigational drug treatment within the 30 days of start of study treatment
* Unsuitable for the study or other chemotherapy determined by investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
No nausea （self report sclae VAS=0）rate in delayed phase (Days2-7) in the first cycle chemotherapy | Day 2-7 in the first chemotherapy cycle(each cycle is 21 days)
  The rate of no nausea on Day 2-7 in the first chemotherapy cycle (each cycle is 21 days).
  The no nausea is defined as score zero with a self-report measure scale,the visual analogue (VAS) scale (0,no symptom, 10, most severely).

SECONDARY OUTCOMES:
No nausea rates （VAS=0）for delayed phases (Days2-7) during 2nd to 4th or 6th chemotherapy cycle,respectively. | Day 2-7 in each chemotherapy cycle (each cycle is 21 days)
  The rates of no nausea on day 2-7 in 2nd-4th or 6th cycle (each cycle is 21 days).
  The no nausea is defined as score zero with a self-report measure scale,the visual analogue (VAS) scale (0,no symptom, 10, most severely).
The complete response rates of vomiting (no emetic episode and no rescue) in acute (Day1),delayed(Day2-7), and overall phase(Day 1-7) during 1st to 4th or 6th cycle, respectively. | Day 1-7 in 4-6 cycles(each cycle is 21 days)
  The rates of no emetic episode and no rescue in acute(Day1),delayed(Day2-7), and overall phase(Day 1-7) during 1st to 4th or 6th cycle, respectively.(each cycle is 21 days). An emetic episode is defined as one occurrence of vomiting or a sequence of occurrences in close succession not relieved by a rest period of at least 1 min; any number of episodes of retching in a 5-minute period; or an episode of retching of , 5 minutes combined with vomiting not relieved in a 1-minute period.
The rate of no anorexia (VAS=0) and score of anorexia (assessed by VAS) in Day1-7 during 1st-4th or 6th cycle chemotherapy | Day 1-7 in each cycle(each cycle is 21 days)
  The rate of no anorexia (VAS=0) and score of anorexia assessed by VAS in multi-cycle chemotherapy. Anorexia score is evaluated with VAS (0,no symptom, 10, most severely)
The score of fatigue by VAS in day1-7 in1st to 4th or 6th chemotherapy cycle,respectively. | Day 1-7 in each cycle(each cycle is 21 days)
  The score of fatigue by self-report scale VAS in day1-7 in1st to 4th or 6th chemotherapy. fatigue is evaluated with self-report scale VAS (0,no symptom, 10, most severely）
The score of sedation(by self-report VAS) in day 1-7 in each cycle | Day 1-7 in each cycle(each cycle is 21 days)
  The score of sedation(by self-report VAS) in day 1-7 in each cycle, respectively.Sedation is evaluated with self-report VAS (0,no symptom, 10, most severely）
Treatment-Related Adverse Events as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 in multi-cycle chemotherapy | Day 1-21 in each cycle(each cycle is 21 days) during 4-6 chemotherapy cycles (each cycle is 21 days)
  Number of participants with Treatment-Related Adverse Events as assessed by CTCAE v4.0, in 4-6 cycles (each cycle is 21 days).
The quality of life scores (evaluated with Functional Living Index-Emesis (FLIE) questionnaire) of patients when receiving multi-cycle chemotherapy | Day 1-8 in each cycle(each cycle is 21 days) during 4-6 chemotherapy cycles.
  The change of quality of life scores from baseline of patients (before chemotherapy) to D8 after chemotherapy in each cycle (each cycle is 21 days). The quality of life are evaluated with Functional Living Index-Emesis (FLIE) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, PhD. M.D., Principal Investigator — China Medical University, China
Locations (29):
- China (29):
  - cancer hospital of Haerbin Medical University, Haerbin, Heilongjiang
  - Siping City Cancer Hospital, Siping, Jilin
  - Anshan Hospital of First Hospital of China Medical University, Anshan, Liaoning
  - Anshan Tumor Hospital, Anshan, Liaoning
  - Central hospital of Dalian, Dalian, Liaoning
  - Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The Fifth Hospital of Dalian City, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Zhuanghe Central Hospital, Dalian, Liaoning
  - Fushun Central Hospital, Fushun, Liaoning
  - General Hospital of Mining Bureau, Fushun, Liaoning
  - Jinzhou Central Hospital, Jinzhou, Liaoning
  - The First Hospital of Liaoning Medical University, Jinzhou, Liaoning
  - Chinese Medicine Hospital of Liaoyang county, Liaoyang, Liaoning
  - Liaoyang Central Hospital, Liaoyang, Liaoning
  - Petrochemical General Hospital of Liaoyang city, Liaoyang, Liaoning
  - Panjin central Hospital, Panjin, Liaoning
  - Chest Hospital of Shenyang City, Shengyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - Liaoning Tumor Hospital & Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - the People'S Hospital, Shenyang, Liaoning
  - Tieling city Central Hospital, Tieling, Liaoning
  - Central Hospital of Anshan City, Anshan
  - Benxi Central Hospital, Benxi
  - Chaoyang Central Hospital, Chaoyang
  - Zhongshan Hospital, Dalian
  - Liaohe Oilfield General Hospital, Panjin

IPD SHARING:
Plan to Share IPD: No